CLINICAL TRIAL: NCT04058457
Title: Deep Brain Stimulation in Parkinson's Disease: Respiratory Testing
Brief Title: DBS and Respiration
Status: Recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Oxford Brookes University (Other)
Responsible Party: Sponsor
Other Study IDs: 256825
Record Dates: First submitted 2019-07-18; First posted 2019-08-15 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; movement disorder; dyspnoea; dyspnea; breathlessness; respiratory
MeSH Terms: conditions — Parkinson Disease; Movement Disorders; Dyspnea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- STN DBS: Patients planned to undergo deep brain stimulation of the subthalamic nucleus
  Interventions: Device: DBS
- GPi DBS: Patients planned to undergo deep brain stimulation of the globus pallidus interna
  Interventions: Device: DBS
- VIM DBS: Patients planned to undergo deep brain stimulation of the ventral intermediate nucleus of thalamus.
  Interventions: Device: DBS

INTERVENTIONS:
Device: DBS — Patients are tested pre-operatively and the post-operatively with their implanted neurostimulators ON and OFF. DBS implantation itself is part of routine care, and not part of the study.

SUMMARY:
Patients referred to neurosurgery routinely and safely undergo deep brain stimulation (DBS) for treatment of neurological conditions, most commonly Parkinson's disease.

The investigators have observed that respiratory problems (breathlessness) sometimes occur subsequent to DBS of the subthalamic nucleus (STN). This study aims to determine whether this is indeed a consequence of STN stimulation. Secondary objectives include identification of the respiratory physiological mediators of any interoceptive neuromodulation observed, changes in daily physical activity and MRI structural connectivity analysis.

DETAILED DESCRIPTION:
A continuous cohort of Parkinson disease patients planned to undergo STN-DBS will be approached to participate in this study (i.e. every patient will be offered participation in the study). Over the same time period other DBS patients (GPi and VIM) will be approached before their implantation procedure to participate as controls/comparators. Participants will all be offered the full study, but will also be free to participate in a smaller number of activities if so chosen.

Patients will be assessed both pre-operatively and post-operatively where they will complete a compound respiratory questionnaire and tests of respiratory interoception and function. Post-operatively, these tests will be carried out with stimulation ON and OFF, the order of which will be randomised between patients.

Data on daily activity will be collected during pre- and post-operative windows, using a wearable pedometer/heart-rate monitor.

Positive findings of respiratory neuromodulation will be correlated between patients with structural connectivity (e.g. STN-insula.) from pre-operative MRI scans.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or female, aged 18 years or above.
* Planned for required DBS surgery
* Fluent in the English language
* For experimental group: diagnosed with Parkinson's disease

Exclusion Criteria:

* Female who is pregnant
* Subject is currently participating in a clinical investigation that includes an active treatment arm which may affect the respiratory system.
* Acute respiratory problem at time of experimental session: e.g. rhinosinusitis, pharyngitis, asthma exacerbation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: STN (Parkinson's disease) GPi (movement disorder, control) VIM (movement disorder, control)
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-07-21 (Estimated); Study Completion 2026-09-21 (Estimated)

PRIMARY OUTCOMES:
Change in breathlessness | Pre-operatively and post-operatively (6-months)
  Dyspnoea questionnaire (D12, MRC)
Change in breathlessness | ON and OFF stimulation between 1 and 6 months after surgery
  Breathlessness ratings (modified-Borg Scale) from experimentally induced breathlessness. 0 = none, 10 maximum. Reported every 15 seconds.

SECONDARY OUTCOMES:
Change in pulmonary function | ON and OFF stimulation between 1 and 6 months after surgery
  Spirometry
Change in airways resistance | ON and OFF stimulation between 1 and 6 months after surgery
  Oscillometry
Change in respiratory muscle strength | ON and OFF stimulation between 1 and 6 months after surgery
  Maximum inspiratory/expiratory pressures
Change in surface electromyography of respiratory muscles | ON and OFF stimulation between 1 and 6 months after surgery
  Signal analysis for evidence of tremor
Change in hypercapnic ventilatory response | ON and OFF stimulation between 1 and 6 months after surgery
  Changes in ventilation from incrementally increased inhaled CO2
Change in breath-hold | ON and OFF stimulation between 1 and 6 months after surgery
  Dyspnoea threshold and breakpoint
Change in daily activity | Pre-operatively (10 days) and post-operatively (10 days, within 6 months of surgery once recovered from surgery and programmed)
  Pedometry
Change in daily activity | Pre-operatively (10 days) and post-operatively (10 days within 6 months of surgery once recovered from surgery and programmed)
  Heart rate
MRI structural connectivity | Pre-operative scan with post-operative analysis through study completion at an average of 1 year
  DTI correlation with respiratory outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Alex Green, FRCS, Principal Investigator — University of Oxford
Locations (1):
- John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom